CLINICAL TRIAL: NCT05936736
Title: 24 Gy in One Fraction Urethral-sparing "High-Dose-Rate Like" Stereotactic Body RadioTherapy for Prostate Cancer: a Single-center Non-randomized Prospective Clinical Study (PRO-FAST)
Brief Title: 24 Gy in One Fraction Urethral-sparing "HDR Like" SBRT for Prostate Cancer
Acronym: PRO-FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Nadia Di Muzio, Prof., IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-FAST
Record Dates: First submitted 2023-06-20; First posted 2023-07-10 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Localized Prostate Carcinoma
Keywords: Prostate Cancer; Single fraction SBRT; Urethral sparing HDR like; PSMA PET/CT; Organ movement; Radiomics
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: According to the optimal design of Simon, 13 pts will be enrolled for the first phase of the study. Hypothesis: the proportion of pts free from acute cumulative G ≥3 toxicity (CTCAE v5.0 scale) 1 month after the end of treatment must be < 85% to suspend treatment and > 95% to consider the treatment as safe. The treatment will be interrupted if G3-G4 toxicities and/or biochemical recurrences are recorded within a month in 2 or more pts, otherwise the study will continue with the second phase enrolling another 52 pts for a total of 65 pts. A single fraction SBRT of 24 Gy with the "urethral sparing HDR like" technique will be delivered. Assuming a minimal drop-out, 5 more pts will be enrolled, thus reaching a total number of 70 pts (65 necessary + 5 for any drop-outs). In the absence of worse subsequent toxicity and with a biochemical control comparable to that in the literature as well as historical treatments of our department, the scheme will be considered as safe and effective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 24 Gy in one fraction, urethral sparing HDR like (Experimental): Patients with localized prostate cancer - negative PSMA PET CT +/- standard staging exams (bone scan, CT, MRI)-enrolled in this study, will be treated to prostate/prostate seminal vesicles (according to the risk group) to a total dose of 24 Gy delivered in 1 fraction, with a urethral sparing HDR like technique. For unfavorable intermediate and high-risk pts, Androgen Deprivation Therapy (ADT) will be prescribed for 6 and 24 months, respectively. The procedure will be performed in just one day, from fiducials implantation to radiation treatment delivery.
  Interventions: Radiation: prostate SBRT

INTERVENTIONS:
Radiation: prostate SBRT — Patients with prostate cancer will be treated with high-dose SBRT to prostate and seminal vesicles, delivered in one fraction, sparing the urethra and generating a dose distribution similar to HDR brachytherapy
  Other Names: ultrahypofractionation; extreme hypofractionation

SUMMARY:
Patients with prostate cancer who are candidates for stereotactic radiotherapy to the prostate and seminal vesicles will undergo staging exams, which will include prostate specific membrane antigen (PSMA) positron emission tomography-computed tomography (PET-CT). If the PET scan is negative and the uroflowmetry is acceptable, the patients will perform the treatment, after fiducial implantation, simulation CT and magnetic resonance (MR), in a single fraction, delivered with a high-dose-rate (HDR)-like urethral sparing technique. In 70 patients, acute and late toxicity, biochemical control, overall survival, cancer specific-survival, and quality of life (through specific questionnaires) will be evaluated.

DETAILED DESCRIPTION:
This is an interventional prospective non-randomised single-center trial that will enroll, 13 patients for the first phase of the study, according to the optimal design of Simon. The hypothesis is that the proportion of patients free from acute cumulative G3-G4 toxicity (Common Terminology Criteria for Adverse Events-CTCAE v5.0 scale) 1 month after the end of treatment must be < 85% to suspend treatment and > 95% to consider the treatment as safe.

The treatment will be interrupted if G3-G4 toxicities and/or biochemical recurrences are recorded within a month in 2 or more patients; otherwise the study will continue with the second phase. Another 52 patients will be added, for a total of 65 patients. The treatment consists in a single fraction of 24 Gy with the "urethral sparing HDR like" technique. Assuming a minimal drop-out, given that the primary endpoint is toxicity one month after treatment, we will enroll 5 more patients in total, thus reaching a total number of 70 patients (65 necessary + 5 for any drop-outs).

In the absence of worse subsequent toxicity, and with biochemical control comparable to that in the literature as well as historical treatments in our Radiation Oncology, the scheme will be considered safe, and the enrollment will continue open label.

Patients with negative lymph nodes and without distant metastases will be enrolled and treated on the prostate/prostate and tumor vesicles (depending on the stage) at a total dose of 24 Gy delivered in a single fraction, sparing the urethra and with a dose distribution similar to high dose rate brachytherapy. Androgen Deprivation Therapy (ADT) will be prescribed according to the guidelines for the stages of the disease.

Short-term cortisone and alpha lytics will be prescribed, for prophylactic purposes. Follow-up visits will be performed at 1, 3, 6,12,18, 24, 36, 48, 60 months with blood tests including prostate specific antigen (PSA) and testosterone (performed every 3 months in the first two years, every 6 months in the next 3 years), imaging, when needed, and quality of life questionnaires: European Organization for Research and Treatment of cancer (EORTC) quality of life questionnaire (QLQ) C30 and QLQ-PR25, International Prostate symptoms score (IPSS), International Index of Erectile Function (IIEF)-5, Expanded Prostate Cancer Index Composite (EPIC)- 26.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of prostate adenocarcinoma, International Society of Urological Pathology (ISUP) grade groups 1-5
* Patients over 18 years of age
* Signed informed consent
* Negative lymph nodes confirmed by imaging (PSMA PET/CT and/or pelvic MRI with and without contrast medium) where recommended by guidelines (intermediate and high risk patients, according to National Comprehensive Cancer Network (NCCN) guidelines) in the previous 3 months
* Clinical M0 (PSMA PET/CT and/or bone scan and/or pelvic MRI with and without contrast medium in suspected patients and unfavorable intermediate and high risk patients, according to NCCN guidelines), in the previous 3 months
* Acceptable uroflowmetry: peak urine flow index (peak flow preferably ≥ 15 ml/s), post voiding residue (PVR) ≤50 cc. If lower, acceptable if, by carrying out 3 months of neoadjuvant hormone therapy + alpha-lytic for the reduction of prostate volume, uroflowmetry is reset to at least ≥ 12 ml/s.
* PS (ECOG) ≤2
* No previous pelvic radiotherapy
* Other conditions necessary for the correct execution of the proposed treatment (ability to fill in the questionnaires for the evaluation of the Quality of Life EORTC QLQ-C30, EORTC QLQ-PR25, IPSS, IIEF-5, EPIC 26)

Exclusion Criteria:

* Serious systemic diseases
* Psychic or other disorders that may prevent the patient from signing the informed consent
* Previous invasive cancer, except skin cancer (excluding melanoma) unless patient free of disease for at least 3 years (e.g. carcinoma in situ of the oral cavity or bladder)
* Lymph node disease (N1)
* Evidence of distant metastases (M1)
* IPSS questionnaire data > 20 points
* Uroflowmetry with maximum basal flow ≤ 11 ml/sec and/or PVR >100 ml
* Concomitant urinary/gastrointestinal inflammatory diseases (e.g. ulcerative colitis, Crohn's disease)
* Overactive bladder
* Impossibility of implantation of fiducials
* Inability or refusal to place bladder catheter for simulation CT and MR
* Inability to perform simulation MRI
* Contraindication for hormonal treatment for patients with unfavorable intermediate, high or very high risk disease
* Non-compliance with dose limits established in the treatment plan

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with prostate
Enrollment: 70 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | one month
  Incidence of acute toxicity of grade 3 or 4 as maximum toxicity value during the radiation treatment or in any case within a month of the end of SBRT, using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 scale (toxicity from 0- patients without toxicity to 5-death from toxicity)

SECONDARY OUTCOMES:
Biochemical control | 5 years (with interim analyzes at 1 and 3 years)
  Biochemical control rate at 1,3 and 5 years by measuring Prostate Specific Antigen-PSA- value which must be below (2+nadir) ng/ml
Biochemical relapse | 5 years (with interim analyzes at 1 and 3 years)
  Biochemical Relapse-Free survival
Local Control | 5 years (with interim analyzes at 1 and 3 years)
  Local Relapse-Free survival
Distant Disease Control | 5 years (with interim analyzes at 1 and 3 years)
  Distant Metastases-Free Survival
Survival | 5 years (with interim analyzes at 1 and 3 years)
  Overall Survival
Subacute Toxicity | 3 months
  Subacute toxicity rated on CTCAE v5.0 scale (see Outcome 1 for details)
Late Toxicity | 5 years (with interim analyzes at 1 and 3 years)
  Late toxicity rated on using CTCAE v5.0 scale (see Outcome 1 for details)
Incidence of Treatment-Emergent Adverse Events as assessed with general quality of life questionnaires | 5 years
  Survey with the questionnaire of European Organisation for Research and Treatment of Cancer (EORTC) Quality of life of cancer patients (QLQ C30) which contains 30 questions on patients' quality of life with answers from 1, lowest grade, to 4, highest grade
Incidence of Treatment-Emergent Adverse Events as assessed with prostate specific quality of life questionnaires | 5 years
  Survey with the questionnaire of European Organisation for Research and Treatment of Cancer (EORTC) Quality of life of prostate cancer patients (QLQ PR25) which contains 25 questions on patients' quality of life with answers from 1, lowest grade, to 4, highest grade
Incidence of Treatment-Emergent Adverse Events as assessed with urinary quality of life questionnaires | 5 years
  Survey with the questionnaire International Prostatic Symptoms Score (IPSS) which has 8 questions with answers rom never (0) to almost every time (5). The score is obtained by summing the answers
Incidence of Treatment-Emergent Adverse Events as assessed with erectile quality of life questionnaires | 5 years
  Survey with the questionnaire IIEF-5 (International Index of Erectile Function). The IIEF-5 score is the sum of the ordinal responses to the 5 items, with higher scores indicating no erectile dysfunction and lower scors indicating severe erectile dysfunction.
Incidence of Treatment-Emergent Adverse Events as assessed with composite quality of life questionnaires | 5 years
  Survey with the questionnaire EPIC-26 (The Expanded Prostate Cancer Index Composite) a questionnaire designed to measure Quality of Life issues in patients with Prostate cancer, through 13 questions with answers from 1 to 5, with 1 indicating the absence of the problem and 5 indicating an important problem. Lower scores indicate a better outcome

OTHER OUTCOMES:
Organ movement | 3 years
  Modeling of organ movements during treatment: Movements of the target and neighboring organs between the treatment fractions and during the treatment will be quantified in millimeters, the median value will be recorded with the range and mean with the standard deviation, and the contributing factors will be identified to find a useful solution
Radiomics | 5 years ( with interim analyzes at 3 years)
  Evaluation of radiomic characteristics: Mathematical extraction of the spatial distribution of signal intensities and pixel interrelationships of medical images of the patients, to quantify textural information resampled according to International Biomarker Standardization Initiative (IBSI).

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Di Muzio, Prof, Study Director — IRCCS San Raffaele Scientific Institute; Andrei Fodor, MD, Study Chair — IRCCS San Raffaele Scientific institute
Locations (1):
- San Raffaele Scientific Institute, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study (anonymized individual participant data) are available on request from the corresponding author to researchers who provide a methodologically sound proposal. Requests made to the corresponding author will be evaluated by the IRCCS San Raffaele Scientific Institute Ethics Committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years after the end of the study
Access Criteria: Request made to PI prof. Nadia Di Muzio or co-PI Dr. Andrei Fodor, approved by Scientific Institute for Research, Hospitalization and Healthcare (IRCCS) San Raffaele Ethics Committee

REFERENCES:
- [Result] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Result] Donovan JL, Hamdy FC, Lane JA, Mason M, Metcalfe C, Walsh E, Blazeby JM, Peters TJ, Holding P, Bonnington S, Lennon T, Bradshaw L, Cooper D, Herbert P, Howson J, Jones A, Lyons N, Salter E, Thompson P, Tidball S, Blaikie J, Gray C, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Davis M, Turner EL, Martin RM, Neal DE; ProtecT Study Group*. Patient-Reported Outcomes after Monitoring, Surgery, or Radiotherapy for Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1425-1437. doi: 10.1056/NEJMoa1606221. Epub 2016 Sep 14. PMID 27626365
- [Result] Prada PJ, Cardenal J, Blanco AG, Anchuelo J, Ferri M, Fernandez G, Arrojo E, Vazquez A, Pacheco M, Fernandez J. High-dose-rate interstitial brachytherapy as monotherapy in one fraction for the treatment of favorable stage prostate cancer: Toxicity and long-term biochemical results. Radiother Oncol. 2016 Jun;119(3):411-6. doi: 10.1016/j.radonc.2016.04.006. Epub 2016 Apr 22. PMID 27118583
- [Result] Prada PJ, Ferri M, Cardenal J, Blanco AG, Anchuelo J, Diaz de Cerio I, Vazquez A, Pacheco M, Raba I, Ruiz S. High-dose-rate interstitial brachytherapy as monotherapy in one fraction of 20.5 Gy for the treatment of localized prostate cancer: Toxicity and 6-year biochemical results. Brachytherapy. 2018 Nov-Dec;17(6):845-851. doi: 10.1016/j.brachy.2018.06.002. Epub 2018 Jul 18. PMID 30030111
- [Result] Pollack A, Zagars GK, Starkschall G, Antolak JA, Lee JJ, Huang E, von Eschenbach AC, Kuban DA, Rosen I. Prostate cancer radiation dose response: results of the M. D. Anderson phase III randomized trial. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1097-105. doi: 10.1016/s0360-3016(02)02829-8. PMID 12128107
- [Result] Kuban DA, Tucker SL, Dong L, Starkschall G, Huang EH, Cheung MR, Lee AK, Pollack A. Long-term results of the M. D. Anderson randomized dose-escalation trial for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):67-74. doi: 10.1016/j.ijrobp.2007.06.054. Epub 2007 Aug 31. PMID 17765406
- [Result] Hall MD, Schultheiss TE, Smith DD, Tseng BP, Wong JY. The impact of increasing dose on overall survival in prostate cancer. Radiat Oncol. 2015 May 21;10:115. doi: 10.1186/s13014-015-0419-3. PMID 25990489
- [Result] Dearnaley D, Syndikus I, Mossop H, Khoo V, Birtle A, Bloomfield D, Graham J, Kirkbride P, Logue J, Malik Z, Money-Kyrle J, O'Sullivan JM, Panades M, Parker C, Patterson H, Scrase C, Staffurth J, Stockdale A, Tremlett J, Bidmead M, Mayles H, Naismith O, South C, Gao A, Cruickshank C, Hassan S, Pugh J, Griffin C, Hall E; CHHiP Investigators. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: 5-year outcomes of the randomised, non-inferiority, phase 3 CHHiP trial. Lancet Oncol. 2016 Aug;17(8):1047-1060. doi: 10.1016/S1470-2045(16)30102-4. Epub 2016 Jun 20. PMID 27339115
- [Result] Catton CN, Lukka H, Gu CS, Martin JM, Supiot S, Chung PWM, Bauman GS, Bahary JP, Ahmed S, Cheung P, Tai KH, Wu JS, Parliament MB, Tsakiridis T, Corbett TB, Tang C, Dayes IS, Warde P, Craig TK, Julian JA, Levine MN. Randomized Trial of a Hypofractionated Radiation Regimen for the Treatment of Localized Prostate Cancer. J Clin Oncol. 2017 Jun 10;35(17):1884-1890. doi: 10.1200/JCO.2016.71.7397. Epub 2017 Mar 15. PMID 28296582
- [Result] Lee WR, Dignam JJ, Amin MB, Bruner DW, Low D, Swanson GP, Shah AB, D'Souza DP, Michalski JM, Dayes IS, Seaward SA, Hall WA, Nguyen PL, Pisansky TM, Faria SL, Chen Y, Koontz BF, Paulus R, Sandler HM. Randomized Phase III Noninferiority Study Comparing Two Radiotherapy Fractionation Schedules in Patients With Low-Risk Prostate Cancer. J Clin Oncol. 2016 Jul 10;34(20):2325-32. doi: 10.1200/JCO.2016.67.0448. Epub 2016 Apr 4. PMID 27044935
- [Result] Fowler JF, Toma-Dasu I, Dasu A. Is the alpha/beta ratio for prostate tumours really low and does it vary with the level of risk at diagnosis? Anticancer Res. 2013 Mar;33(3):1009-11. PMID 23482774
- [Result] Miralbell R, Roberts SA, Zubizarreta E, Hendry JH. Dose-fractionation sensitivity of prostate cancer deduced from radiotherapy outcomes of 5,969 patients in seven international institutional datasets: alpha/beta = 1.4 (0.9-2.2) Gy. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):e17-24. doi: 10.1016/j.ijrobp.2010.10.075. Epub 2011 Feb 15. PMID 21324610
- [Result] Dasu A, Toma-Dasu I. Prostate alpha/beta revisited -- an analysis of clinical results from 14 168 patients. Acta Oncol. 2012 Nov;51(8):963-74. doi: 10.3109/0284186X.2012.719635. Epub 2012 Sep 12. PMID 22966812
- [Result] Katz AJ, Santoro M, Diblasio F, Ashley R. Stereotactic body radiotherapy for localized prostate cancer: disease control and quality of life at 6 years. Radiat Oncol. 2013 May 13;8:118. doi: 10.1186/1748-717X-8-118. PMID 23668632
- [Result] King CR, Freeman D, Kaplan I, Fuller D, Bolzicco G, Collins S, Meier R, Wang J, Kupelian P, Steinberg M, Katz A. Stereotactic body radiotherapy for localized prostate cancer: pooled analysis from a multi-institutional consortium of prospective phase II trials. Radiother Oncol. 2013 Nov;109(2):217-21. doi: 10.1016/j.radonc.2013.08.030. Epub 2013 Sep 20. PMID 24060175
- [Result] Fuller DB, Falchook AD, Crabtree T, Kane BL, Medbery CA, Underhill K, Gray JR, Peddada A, Chen RC. Phase 2 Multicenter Trial of Heterogeneous-dosing Stereotactic Body Radiotherapy for Low- and Intermediate-risk Prostate Cancer: 5-year Outcomes. Eur Urol Oncol. 2018 Dec;1(6):540-547. doi: 10.1016/j.euo.2018.06.013. Epub 2018 Jul 25. PMID 31158102
- [Result] Kishan AU, Dang A, Katz AJ, Mantz CA, Collins SP, Aghdam N, Chu FI, Kaplan ID, Appelbaum L, Fuller DB, Meier RM, Loblaw DA, Cheung P, Pham HT, Shaverdian N, Jiang N, Yuan Y, Bagshaw H, Prionas N, Buyyounouski MK, Spratt DE, Linson PW, Hong RL, Nickols NG, Steinberg ML, Kupelian PA, King CR. Long-term Outcomes of Stereotactic Body Radiotherapy for Low-Risk and Intermediate-Risk Prostate Cancer. JAMA Netw Open. 2019 Feb 1;2(2):e188006. doi: 10.1001/jamanetworkopen.2018.8006. PMID 30735235
- [Result] Jackson WC, Silva J, Hartman HE, Dess RT, Kishan AU, Beeler WH, Gharzai LA, Jaworski EM, Mehra R, Hearn JWD, Morgan TM, Salami SS, Cooperberg MR, Mahal BA, Soni PD, Kaffenberger S, Nguyen PL, Desai N, Feng FY, Zumsteg ZS, Spratt DE. Stereotactic Body Radiation Therapy for Localized Prostate Cancer: A Systematic Review and Meta-Analysis of Over 6,000 Patients Treated On Prospective Studies. Int J Radiat Oncol Biol Phys. 2019 Jul 15;104(4):778-789. doi: 10.1016/j.ijrobp.2019.03.051. Epub 2019 Apr 6. PMID 30959121
- [Result] Widmark A, Gunnlaugsson A, Beckman L, Thellenberg-Karlsson C, Hoyer M, Lagerlund M, Kindblom J, Ginman C, Johansson B, Bjornlinger K, Seke M, Agrup M, Fransson P, Tavelin B, Norman D, Zackrisson B, Anderson H, Kjellen E, Franzen L, Nilsson P. Ultra-hypofractionated versus conventionally fractionated radiotherapy for prostate cancer: 5-year outcomes of the HYPO-RT-PC randomised, non-inferiority, phase 3 trial. Lancet. 2019 Aug 3;394(10196):385-395. doi: 10.1016/S0140-6736(19)31131-6. Epub 2019 Jun 18. PMID 31227373
- [Result] Brand DH, Tree AC, Ostler P, van der Voet H, Loblaw A, Chu W, Ford D, Tolan S, Jain S, Martin A, Staffurth J, Camilleri P, Kancherla K, Frew J, Chan A, Dayes IS, Henderson D, Brown S, Cruickshank C, Burnett S, Duffton A, Griffin C, Hinder V, Morrison K, Naismith O, Hall E, van As N; PACE Trial Investigators. Intensity-modulated fractionated radiotherapy versus stereotactic body radiotherapy for prostate cancer (PACE-B): acute toxicity findings from an international, randomised, open-label, phase 3, non-inferiority trial. Lancet Oncol. 2019 Nov;20(11):1531-1543. doi: 10.1016/S1470-2045(19)30569-8. Epub 2019 Sep 17. PMID 31540791
- [Result] Siddiqui ZA, Gustafson GS, Ye H, Martinez AA, Mitchell B, Sebastian E, Limbacher A, Krauss DJ. Five-Year Outcomes of a Single-Institution Prospective Trial of 19-Gy Single-Fraction High-Dose-Rate Brachytherapy for Low- and Intermediate-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2019 Aug 1;104(5):1038-1044. doi: 10.1016/j.ijrobp.2019.02.010. Epub 2019 Feb 13. PMID 30771408
- [Result] Armstrong S, Tsang Y, Lowe G, Tharmalingam H, Alonzi R, Ostler P, Hughes R, Hoskin P. Dosimetry of local failure with single dose 19 Gy high-dose-rate brachytherapy for prostate cancer. Radiother Oncol. 2021 Apr;157:93-98. doi: 10.1016/j.radonc.2021.01.006. Epub 2021 Jan 23. PMID 33493500
- [Result] Greco C, Pares O, Pimentel N, Louro V, Santiago I, Vieira S, Stroom J, Mateus D, Soares A, Marques J, Freitas E, Coelho G, Seixas M, Lopez-Beltran A, Fuks Z. Safety and Efficacy of Virtual Prostatectomy With Single-Dose Radiotherapy in Patients With Intermediate-Risk Prostate Cancer: Results From the PROSINT Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 May 1;7(5):700-708. doi: 10.1001/jamaoncol.2021.0039. PMID 33704378
- [Result] Zelefsky MJ, Yamada Y, Greco C, Lis E, Schoder H, Lobaugh S, Zhang Z, Braunstein S, Bilsky MH, Powell SN, Kolesnick R, Fuks Z. Phase 3 Multi-Center, Prospective, Randomized Trial Comparing Single-Dose 24 Gy Radiation Therapy to a 3-Fraction SBRT Regimen in the Treatment of Oligometastatic Cancer. Int J Radiat Oncol Biol Phys. 2021 Jul 1;110(3):672-679. doi: 10.1016/j.ijrobp.2021.01.004. Epub 2021 Jan 8. PMID 33422612
- [Result] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Derived] Fodor A, Giannini L, Torrisi M, Brombin C, Broggi S, Losa A, Maga T, Mellone R, Martinenghi C, Tummineri R, Mangili P, Deantoni CL, Tudda A, Castriconi R, Rancoita PMV, Di Serio MS, Gaboardi F, Fiorino C, Del Vecchio A, Chiti A, De Cobelli F, Di Muzio N. Comprehensive one-day management of prostate cancer patients: PRO-FAST single-fraction ablative, urethral-sparing, HDR-like, robotic SBRT. Radiat Oncol. 2025 Aug 27;20(1):134. doi: 10.1186/s13014-025-02713-9. PMID 40866948